CLINICAL TRIAL: NCT01478490
Title: An Open Label, One-sequence, Parallel Study to Compare the Single Dose Pharmacokinetics of YM178 in Healthy Poor or Extensive Metabolisers for CYP2D6 and to Assess the Effect of Multiple Doses of YM178 on the Metabolism of the Model Substrate Metoprolol
Brief Title: To Compare Blood and Urine Concentrations of Mirabegron (YM178) in Healthy Poor or Extensive Metabolizers for CYP2D6 and to Assess the Effect of Mirabegron on the Metabolism of Metoprolol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-005
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacokinetics of Mirabegron; Healthy Subjects
Keywords: Pharmacokinetics,; Mirabegron; Metoprolol; CYP2D6; Phase 1
MeSH Terms: interventions — mirabegron; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Arm 1A (Experimental): mirabegron, poor metabolizers
  Interventions: Drug: mirabegron
- Treatment Arm 1B (Experimental): mirabegron, extensive metabolizers
  Interventions: Drug: mirabegron
- Treatment Arm 2 (Experimental): mirabegron/metoprolol
  Interventions: Drug: mirabegron; Drug: metoprolol

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178
Drug: metoprolol — oral
  Arms: Treatment Arm 2

SUMMARY:
The study aims to compare blood and urine concentrations of mirabegron (YM178) in healthy poor or extensive metabolizers for CYP2D6 and to evaluate if blood levels of metoprolol change whilst being dosed at the same time with daily miragebron.

DETAILED DESCRIPTION:
The study is an open label, single center study. All subjects are genotyped for CYP2D6 before the study. Genotype expression is confirmed by dextromethorphan phenotyping.

Part I: The pharmacokinetic profile of a single dose of YM178 is compared in 8 healthy male subjects genotyped and phenotyped as poor metaboliser (PM) for CYP2D6 and in 8 healthy male subjects genotyped and phenotyped as extensive metaboliser (EM) for CYP2D6.

Part II: The effect of YM178 on the model substrate of CYP2D6 metoprolol is evaluated, using a cross-over design, in 12 healthy male subjects genotyped and phenotyped as EM for CYP2D6.

ELIGIBILITY:
Inclusion Criteria:

For Part I:

* Subject genotyped and phenotyped for CYP2D6
* Body weight between 60 and 100 kg and Body Mass Index less than or equal to 30 kg/m2

For Part II:

* Subject genotyped and phenotyped as extensive metaboliser for CYP2D6
* Body weight between 60 and 100 kg and Body Mass Index less than or equal to 30 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to β-adrenergic receptor agonists or constituents of the formulations used
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug
* Any clinically significant history of upper gastrointestinal symptoms (such as nausea, vomiting, abdominal discomfort or upset, or heartburn) in the 4 weeks prior to admission to the Research Unit
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* QTc intervals of >430 msec
* Abnormal pulse rate measurement (<40 or >90 bpm) taken by manual counting at the pre-study visit after subject has been resting in supine position for 5 min
* Abnormal blood pressure measurements taken at the pre-study visit after subject has been resting in supine position for 5 min as follows: systolic blood pressure <95 or >160 mmHg; diastolic blood pressure <40 or >95 mmHg
* Positive orthostatic test at screening i.e. any symptoms of dizziness, light-headedness etc. and/or a fall of ≥ 20 mmHg in systolic blood pressure after 2 min standing (preceded by 5 min. supine rest) and/or an increase in pulse rate of ≥ 20 bpm
* Regular use of any prescribed or OTC drugs except paracetamol up to 3 g/day, in the 4 weeks prior to admission to the Research Unit OR any use of such drugs in the 2 weeks prior to admission to the Research Unit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-09; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of mirabegron assessed by plasma concentration | Pre-dose until 72 hours after dosing
  Primary outcome measure for Part 1

SECONDARY OUTCOMES:
Pharmacokinetics of metoprolol assessed by plasma concentration | Pre-dose until 48 hours after dosing
  Primary outcome measure for Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — Pharma Bio-Research Group B.V., Zuidlaren, The Netherlands
Locations (1):
- PRA International (former Pharma Bio-Research), Zuidlaren, Netherlands

REFERENCES:
- [Background] Krauwinkel W, Dickinson J, Schaddelee M, Meijer J, Tretter R, van de Wetering J, Strabach G, van Gelderen M. The effect of mirabegron, a potent and selective beta3-adrenoceptor agonist, on the pharmacokinetics of CYP2D6 substrates desipramine and metoprolol. Eur J Drug Metab Pharmacokinet. 2014 Mar;39(1):43-52. doi: 10.1007/s13318-013-0133-1. Epub 2013 Jun 1. PMID 23728524